CLINICAL TRIAL: NCT02816398
Title: Vessel-Select Catheter System Feasibility Clinical Trial
Brief Title: Catheter System Feasibility Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Collaborators: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-0012-01
Record Dates: First submitted 2016-06-23; First posted 2016-06-28 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2016-06

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Interventional use of experimental Ellipsys catheter system for percutaneous creation of an arteriovenous fistula
  Interventions: Device: Percutaneous creation of an arteriovenous fistula

INTERVENTIONS:
Device: Percutaneous creation of an arteriovenous fistula — Use of catheter system for percutaneous creation of an arteriovenous fistula

SUMMARY:
Feasibility clinical study to evaluate the safety and effectiveness of the catheter system for the percutaneous creation of an arteriovenous fistula for patients with end stage renal disease requiring dialysis access.

ELIGIBILITY:
Inclusion Criteria:

* Patients deemed medically eligible for AV fistula creation per institutional guidelines and/or clinical judgment
* Patients diagnosed with chronic kidney disease classification stage IV or V
* Adequate quality vein >= 2 mm with confirmed clinically significant outflow based on pre-operative assessment
* Adequate quality radial artery >= 2 mm based on pre-operative assessment
* Adequate collateral arterial perfusion
* Radial artery-adjacent vein proximity < = 1.5 mm
* Able to provide informed consent
* Able to travel to institution for follow up examination
* Able to intraoperatively place an .014" guidewire in artery

Exclusion Criteria:

* Suspected skin disease
* Immunocompromised patients (e.g. HIV positive)
* Edema of extremities
* Current diagnosis of carcinoma
* Pregnancy or currently breast feeding
* Diagnosed hypercoaguable state
* Active infection
* Evidence of vascular disease at target site
* Pre-existing vascular disease that could confound study results
* Vessel tortuosity or spasm preventing placement of .014" guidewire

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 26
Completed | 12
Not Completed | 14
Not completed — Death | 5
Not completed — Lack of Efficacy | 8
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 26
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sufficient Patency for Clinical Access
Description: Arteriovenous fistula is patent as determined by auscultation or ultrasound and eligible for maturation assistance to achieve clinical access flow rate.
Time Frame: 6 weeks
Population: Patency at 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 26
Participants | 20

2. Primary Outcome: Number of Patients Achieving Dialysis Access
Description: Arteriovenous fistula is mature and patient has started dialysis using the fistula
Time Frame: 6 weeks
Population: Patients on dialysis at 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 26
Participants | 1

3. Primary Outcome: Number of Patients on Dialysis Using the Arteriovenous Fistula or Has Adequate Access Flow Rate to Allow Dialysis
Description: Arteriovenous fistula is mature or has achieved a minimum clinically acceptable access flow rate as determined by doppler ultrasound assessment to support dialysis
Time Frame: 3 months
Population: Patients on dialysis or achieved suitable access flow rate
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 26
Participants | 20

4. Secondary Outcome: Number of Patients Requiring Additional Interventions to Achieve Maturation and Dialysis Access
Description: The number of patients requiring additional interventions to achieve maturation and initiation of dialysis.
Time Frame: 12 weeks
Population: Number of additional interventions to achieve suitability for dialysis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 26
Participants | 23

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of 6 months from index procedure through arteriovenous fistula maturation
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 9/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=23)
Death (General disorders) | 5 (5) — Deaths during study duration. None related to treatment procedure
Hematoma (Blood and lymphatic system disorders) | 1 (1) — Hematoma associated with procedure
Acute thrombosis (Vascular disorders) | 3 (3) — Acute thrombosis of anastomosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No